CLINICAL TRIAL: NCT00129090
Title: A Randomized Phase III Study to Compare Conventional Chemotherapy (CHOEP-14) + Rituximab vs High-dose Chemotherapy Followed by Autologous Stem Cell Transplantation (Mega-CHOEP-21) + Rituximab in Younger Patients With Aggressive NHL
Brief Title: Mega-CHOEP: Conventional Chemo Vs HD Chemo Followed by Auto SCT in Younger Pts With Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL 2002-1
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Non-Hodgkin's Lymphoma (NHL)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CHOEP14 with 12x Rituximab (Experimental): 8 cycles of standard CHOP with etoposide in 14-day intervals. Patients with CD20+ lymphoma receive 12 doses of Rituximab (day 0,1,4,8 of cycle 1, day 1 and 8 of cycle 2, day1 of cycle 3-8 )
  Interventions: Drug: R-CHOEP 14 with 12x Rituximab

INTERVENTIONS:
Drug: R-CHOEP 14 with 12x Rituximab — after amendment 3 patients receive 4x 375mg/m2 in cycle 1 (day 0,1,4,8), 2x 375/m2 in cycle 2 (day1,8) and 1x 375mg/m2 cycle 3-8 (day 1 of each cycle)
  Other Names: 12 x Rituximab with 8 cycles of standard CHOEP-14

SUMMARY:
According to amendment 3 this study addresses the question if intensification of administration of rituximab in standard treatment for patients with newly diagnosed aggressive B-Non Hodgkin Lymphoma (B-NHL) and high risk (aaIPI 2 or 3) results in a better time to treatment failure (TTTF)

DETAILED DESCRIPTION:
This study was primarily designed to compare aggressive conventional chemotherapy with a repetitive high-dose (HD) therapy program using identical, effective drugs at highest possible dose and dose intensity with/without addition of rituximab (initially 4 treatment arms). In 2004 the first amendment had to be added in order to close two treatment arms without rituximab due to recent data revealing a significant advantage for rituximab-treated patients with CD20+lymphoma.

A planned interim analysis in 2010 revealed inferiority of the high-dose treatment thus in the 2nd amendment the high-dose arm was closed and additionally the rituximab frequency was raised from 6 to 12 administrations as recent publications gave hint for advantage. The last amendment was added in 2010 to adjust for delayed recruitment mainly due to organisation problems.

As the high-dose arm was closed only CD20+ B-lymphoma were included past amendment 2.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Risk group International Prognostic Index (IPI) 2 and 3 (age adjusted)
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-3
* Patient's written informed consent
* Aggressive non-Hodgkin's lymphoma with CD20+ histology

Exclusion Criteria:

* Already initiated lymphoma therapy
* Serious accompanying disorder or impaired organ function
* Bone marrow involvement > 25%
* Known hypersensibility to the medications to be used
* Known HIV-positivity
* Active hepatitis infection
* Suspicion that patient compliance will be poor
* Simultaneous participation in other trials
* Prior chemo- or radiotherapy for previous disorder
* Other concomitant tumour disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2003-03; Primary Completion 2014-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
time to treatment failure | 3 years after study inclusion
  At 3 year follow up rate of treatments and time to treatment failure will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Schmitz, Prof., Principal Investigator — German High-Grade Non-Hodgkin's Lymphoma Study Group
Locations (1):
- AK St. Georg, Hamburg, Germany

REFERENCES:
- [Derived] Oertel M, Ziepert M, Frontzek F, Nacke N, Altmann B, Nickelsen M, Glass B, Poeschel V, Ruebe C, Lenz G, Schmitz N, Eich HT. Radiotherapy in younger patients with advanced aggressive B-cell lymphoma-long-term results from the phase 3 R-MegaCHOEP trial. Leukemia. 2024 May;38(5):1099-1106. doi: 10.1038/s41375-024-02231-9. Epub 2024 Mar 27. PMID 38538861
- [Derived] Frontzek F, Ziepert M, Nickelsen M, Altmann B, Glass B, Haenel M, Truemper L, Held G, Bentz M, Borchmann P, Dreyling M, Viardot A, Kroschinsky FP, Metzner B, Staiger AM, Horn H, Ott G, Rosenwald A, Loeffler M, Lenz G, Schmitz N. Rituximab plus high-dose chemotherapy (MegaCHOEP) or conventional chemotherapy (CHOEP-14) in young, high-risk patients with aggressive B-cell lymphoma: 10-year follow-up of a randomised, open-label, phase 3 trial. Lancet Haematol. 2021 Apr;8(4):e267-e277. doi: 10.1016/S2352-3026(21)00022-3. Epub 2021 Mar 2. PMID 33667420
- [Derived] Schmitz N, Nickelsen M, Ziepert M, Haenel M, Borchmann P, Schmidt C, Viardot A, Bentz M, Peter N, Ehninger G, Doelken G, Ruebe C, Truemper L, Rosenwald A, Pfreundschuh M, Loeffler M, Glass B; German High-Grade Lymphoma Study Group (DSHNHL). Conventional chemotherapy (CHOEP-14) with rituximab or high-dose chemotherapy (MegaCHOEP) with rituximab for young, high-risk patients with aggressive B-cell lymphoma: an open-label, randomised, phase 3 trial (DSHNHL 2002-1). Lancet Oncol. 2012 Dec;13(12):1250-9. doi: 10.1016/S1470-2045(12)70481-3. Epub 2012 Nov 16. PMID 23168367